CLINICAL TRIAL: NCT00489879
Title: Efficacy of Mobile Health Care System in Patients With Type 2 Diabets and Hypertension
Brief Title: Management of Patients With Type 2 Diabetes and Hypertension Using Mobile Health Care System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University (Other)
Responsible Party: Kyung Mook Choi, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Seoul R&BD Program
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Diabetes; Hypertension; Obesity
Keywords: Mobile Health Units; Chronic Disease
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Obesity; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Mobile Health Care System (DrUB)

SUMMARY:
The purpose of this study is to determine whether cellular phone based health care system is effective in the treatment of diabetes and hypertension.

DETAILED DESCRIPTION:
Diabetes care is facilitated by a patient's being engaged in a self-management program with the advice and counsel of physicians, but many diabetic patients can not receive the continous monitoing and advice from his physician in their every day life. It is very difficult to keep up life style modification in their real life.

Few studies have examined the effects of cellular phone based intervention that provide an interactive component daily. Our goal is to test the hypothesis that diabetes and hypertension management using cellular phone based health care system would result in significant improvement of blood glucose and blood pressure level.

ELIGIBILITY:
Inclusion Criteria:

* type II diabetes using only oral hypoglycemic agents
* 7% < HbA1c < 10%
* systolic blood pressure > 130 or diastolic blood pressure > 80
* BMI > 23
* 20 < age < 75

Exclusion Criteria:

* type I diabetes or type II diabtes using insulin treatment
* liver, renal or heart disease
* recent change (within 1 month) in the type or dosage of anti-diabetic agent, anti-hypertensive medication

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2007-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
HbA1c, fasting blood glucose level, Weight change, Blood pressure level in the morning, lipid profiles | baseline, 3months later

SECONDARY OUTCOMES:
exercise time during one week, self reported change in dietary habit, fat consumption ratio | baseline, 3months later

CONTACTS AND LOCATIONS:
Overall Officials: Kyung M Choi, MD, Principal Investigator — Department of Internal Medicine, Korea University College of Medicine
Locations (1):
- Department of Internal Medicine, Korea University College of Medicine, Seoul, VD, South Korea

REFERENCES:
- [Background] Kwon HS, Cho JH, Kim HS, Song BR, Ko SH, Lee JM, Kim SR, Chang SA, Kim HS, Cha BY, Lee KW, Son HY, Lee JH, Lee WC, Yoon KH. Establishment of blood glucose monitoring system using the internet. Diabetes Care. 2004 Feb;27(2):478-83. doi: 10.2337/diacare.27.2.478. PMID 14747232